CLINICAL TRIAL: NCT04405635
Title: Quantifying Digital Behavior on Smart Phones - Data From Stroke Survivors
Acronym: QuantStroke
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Aarhus (Other)
Collaborators: Leiden University (Other); Carlsberg Foundation (Unknown)
Responsible Party: Sponsor
Other Study IDs: 614731
Record Dates: First submitted 2020-05-26; First posted 2020-05-28 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-12

CONDITIONS: Stroke
Keywords: Stroke, digital behavior, health-related quality of life, cognitive function
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention or exposure — No intervention or exposure

SUMMARY:
In this study, we want to continuously record the interaction of 50 stroke survivors with their smartphones during the first 3 months after discharge. The linkage of smart phone use to function and quality of life will be assessed with standardized outcome measures at defined time points.

DETAILED DESCRIPTION:
People with stroke are among the most relevant target groups for unobtrusive monitoring. Worldwide, stroke is the second most frequent cause for lasting disability and causes a substantial burden for the individual, caregivers and society. Thanks to improved treatment, many stroke survivors can be discharged to their homes. However, many have to live with disabilities and are prone to declining function, cognitive impairment and depression. With the acquired data, we want to create a database where digital behavior is analyzed with advanced computational methods. In collaboration with the Department of Cognitive Psychology, University of Leiden, Netherlands, these data will be used to discover specific features for different health issues and to develop tools for the early detection of functional decline for different populations.

ELIGIBILITY:
Inclusion Criteria:

* New or recurrent stroke, admitted to rehabilitation, discharge to own home
* Owns an Android smart phone
* Smart phone is used by the patient only

Exclusion Criteria:

* Severe cognitive impairments and / or psychiatric and behavioral conditions that interfere with compliance.
* Not able to provide informed consent
* Discharge to nursing homes or other care facilities

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We want to include a broad range of patients with stroke, incuding both ischemic and hemorrhagic strokes and different impairments due to stroke. Patients are recruited at two wards specialized in neurorehabilitation around 1 week before discharge to their home.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-05-30 (Actual); Primary Completion 2024-07-28 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Different parameters of digital behavior | Continuously throughout the 90 days of monitoring
  Number of interactions with the smart phone, tapping speed, typing speed, social media use

SECONDARY OUTCOMES:
EQ5D | Once a week during 12 weeks
  Health related quality of life, 5 point subscale, Index values of 0-1 (better), EQ5D VAS 0-100 (better)
Mini MoCA | 3 times in three months, after 4, 8 and 12 weeks
  Montreal Cognitive Assessment, cognitive function, scale 0-15 (better)
SF-36 | 3 times in three months, after 4, 8 and 12 weeks
  Health related quality of life, 0-100 (better)
Stroke Specific Quality of Life Questionnaire - short version | 3 times in three months, after 4, 8 and 12 weeks
  Stroke related quality of life, 12-60 (better)

OTHER OUTCOMES:
Health today | Every day throughout 90 days
  One question about subjective health, VAS 0-100 (better)

CONTACTS AND LOCATIONS:
Overall Officials: Iris C. Brunner, PhD, Principal Investigator — Aarhus University, Hammel Neurocenter
Locations (1):
- Hammel Neurorehabilitation Centre and University Research Clinic, Hammel, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
Processed smartphone behavioral data and the associated processing codes will be made available upon publication and corresponding release in data repositories.